CLINICAL TRIAL: NCT06327009
Title: Effect of Ramadan Fasting on Kidney Function and Proteinuria in Patients With Glomerulonephritis: a Prospective Observational Clinical Trial
Brief Title: Effect of Ramadan Fasting on Kidney Function and Proteinuria in Patients With Glomerulonephritis
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, assistant professor, Alexandria University
Other Study IDs: fasting ramadan in GN patients
Record Dates: First submitted 2024-03-12; First posted 2024-03-25 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Fasting Ramadan
Keywords: fasting ramadan; glomerulonephritis; kidney functions
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fasting: 100 patients who decided to fast the month of ramadan.
  Interventions: Behavioral: fasting month of ramadan

INTERVENTIONS:
Behavioral: fasting month of ramadan — 100 patients with glomerulonephritis who decided to fast month of ramadan

SUMMARY:
This research aims to assess effects of ramadan fasting on kidney function and proteinuria in patients with glomerulonephritis.

DETAILED DESCRIPTION:
Fasting from sunrise to sunset during the Islamic holy month of Ramadan is one of the five pillars of the Islamic faith. Duration of the fasting ranges from 10 to 18 hours per day according to the geographic location and the season. Although people with chronic illnesses are exempted from fasting according to Islamic beliefs, many patients insist on fasting against medical advice. Through the last three decades many reports studied the potential risks and benefits of fasting Ramadan in regular hemodialysis (HD) patients. Target points of investigation were different. Most of them were focusing on the electrolytes and nutritional changes. Fewer reports tested the mortality rate. In a multicenter observational study, 2055 Egyptian patients from 25 HD units were studied for frequency of fasting in Ramadan and the possible effect of fasting on clinical and biochemical variables. The investigators concluded that nearly 47% of the study patients fasted at least few days of Ramadan. They recommended that HD patients should be encouraged to discuss the option of fasting in Ramadan with their HD staff who might be able to give advice on whether to allow them to fast in days off dialysis with special precautions regarding associated comorbidities, especially diabetes and coronary artery disease. Most of the studies focused on the effects of fasting the month of Ramadan in CKD and hemodialysis patients, but no research assessed these effects specifically in patients with glomerulonephritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven glomerulonephritis with eGFR ≥ 30 ml/min for more than 3 months (exception is nephrotic patients with positive anti-PLA2R indicative of primary membranous).

Exclusion Criteria:

* Patients with medical contraindications for fasting.
* Patients with eGFR < 30 ml/min.
* Patients with acute cardiovascular disease.
* uncontrolled diabetes mellitus.
* active or chronic inflammatory disease.
* Acute liver disease.
* Pregnancy.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: one hundred patients with biopsy proven glomerulonephritis for more than 3 months from different centers in Egypt will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Change in kidney function | 4 weeks (month of ramadan)
  By assessing change in eGFR
Change in proteinuria | 4 weeks (month of ramadan)
  By assessing change in protein to creatinine ratio in urine

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — assistant professor; kariem M salem, MD, Study Chair — lecturer
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sahin SB, Ayaz T, Ozyurt N, Ilkkilic K, Kirvar A, Sezgin H. The impact of fasting during Ramadan on the glycemic control of patients with type 2 diabetes mellitus. Exp Clin Endocrinol Diabetes. 2013 Oct;121(9):531-4. doi: 10.1055/s-0033-1347247. Epub 2013 Aug 9. PMID 23934679
- [Background] Megahed AF, El-Kannishy G, Sayed-Ahmed N. Status of fasting in Ramadan of chronic hemodialysis patients all over Egypt: A multicenter observational study. Saudi J Kidney Dis Transpl. 2019 Mar-Apr;30(2):339-349. doi: 10.4103/1319-2442.256841. PMID 31031370